CLINICAL TRIAL: NCT07330557
Title: Effect of the Labour Hopscotch Method on the Labor Process and Maternal Satisfaction: A Randomized Controlled Trial
Brief Title: The Effect Of The Labour Hopscotch On The Birth Process And Satisfaction
Acronym: Labor Hopscotc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Pirozhan, doctoral student, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/46; 2023/46 (Other: Adnan Menderes University Faculty of Health Sciences)
Record Dates: First submitted 2025-12-08; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Labor Duration; Labor Bain; and Birth Satisfaction During Physiologic Vaginal Birth
Keywords: Labor hopscotch; physiologic vaginal birth; labor pain; labor duration,; birth satisfaction; non-pharmacological intrapartum care
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: A parallel design was chosen to compare the effects of the labor hopscotch program with standard intrapartum care. Participants are randomly assigned to either the intervention or control group, and outcomes are measured concurrently in both groups.
Who Masked: Participant
Masking Description: No parties are masked in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor Hopscotch Program Group (Experimental): Participants undergo the Labor Hopscotch Exercise Program during the first stage of labor. This program is a non-pharmacological, behavioral intervention that encourages active movement. The exercises aim to shorten labor duration, reduce pain, and increase birth satisfaction. The program is performed under the supervision of trained healthcare professionals and provides ongoing intrapartum support.
  Interventions: Behavioral: Labor Hopscotch Exercise Program Group; Other: Standard Intrapartum Care
- Standard Intrapartum Care Group → Control (Other): Participants received standard intrapartum care. This intervention included routine birth practices and care procedures. This group, which did not include any special exercises or additional interventions, served as the control group.
  Interventions: Behavioral: Labor Hopscotch Exercise Program Group; Other: Standard Intrapartum Care

INTERVENTIONS:
Behavioral: Labor Hopscotch Exercise Program Group — Throughout labor, active positions, movements, breathing exercises, and recordings are utilized, along with the hopscotch steps.
  Guided by a trained midwife/healthcare professional.
  Applied throughout the latent and active phases.
  Purpose: To reduce pain, facilitate labor progression, and minimize interventions.
Other: Standard Intrapartum Care — The institution's routine standard maternity care protocol
  Nonpharmacological or pharmacological comfort measures per standard care
  Includes routine clinical practices of healthcare professionals
  Hopscotch program is not implemented

SUMMARY:
This study is designed to evaluate the effect of the Labor Hopscotch exercise on the birth process and maternal satisfaction. The study will be conducted as a randomized controlled trial at a tertiary-level maternity unit. Eligible pregnant women will be recruited during the active phase of labor and randomly assigned to either the intervention group or the control group.

Participants in the intervention group will receive the Labor Hopscotch exercise program during labor in addition to standard intrapartum care. The control group will receive standard intrapartum care only. The Labor Hopscotch exercise program consists of structured physical movements adapted to the stages of labor and is implemented under the supervision of trained healthcare professionals.

Data will be collected using standardized data collection forms, obstetric records, and validated measurement tools. Information related to sociodemographic characteristics, obstetric history, labor characteristics, and maternal experiences during labor will be recorded. The study is conducted in accordance with ethical principles and relevant institutional guidelines.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of the Labor Hopscotch exercise on the labor process and maternal experience. The study is designed as a randomized controlled trial including eligible pregnant women. Participants will be allocated to an intervention group or a control group, and predefined outcomes will be assessed using standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women with cervical dilation between 3cm and 5cm, expected to have a vaginal delivery and admitted to the delivery room,
* Pregnant women aged 18-35,
* Pregnant women with gestational age between 37-42 weeks,
* Able to speak and understand Turkish, and
* At least primary school graduates (as the scales will be completed using the self-report method) will be included.
* Pregnant women without a history of mental or physical health problems,
* Pregnant women without a history of high-risk pregnancy.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — • Primiparous pregnant women
Enrollment: 110 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Maternal Satisfaction Score Measured by a Validated Satisfaction Scale | Within 24 hours postpartum
  Maternal satisfaction will be assessed using a validated satisfaction scale. Total scores will be calculated according to the scale guidelines, with higher scores indicating greater maternal satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Kadın ve Çocuk Hastalıkları Hastanesi, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to qualified researchers upon reasonable request after publication of the main study results. Data will be shared through a secure data repository, following ethical and privacy regulations.

REFERENCES:
- [Result] Carroll L, Thompson S, Coughlan B, McCreery T, Murphy A, Doherty J, Sheehy L, Cronin M, Brosnan M, O'Brien D. 'Labour Hopscotch': Women's evaluation of using the steps during labor. Eur J Midwifery. 2022 Sep 9;6:59. doi: 10.18332/ejm/152492. eCollection 2022. PMID 36132188